CLINICAL TRIAL: NCT01723397
Title: Effect of Nasaleze on the Early Reaction to Nasal Challenge With Allergen
Brief Title: Effect of Nasaleze on Nasal Challenge With Allergen
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-1252
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Allergens

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasaleze spray (Active Comparator): Nasaleze spray 1 puff via "spray device" in each nostril 3 times daily for 1 week followed by allergen challenge
  Interventions: Drug: Nasaleze Spray; Biological: Allergen
- Placebo spray (Placebo Comparator): Placebo spray 1 puff via "spray device" in each nostril 3 times daily for 1 week followed by allergen challenge
  Interventions: Other: Placebo spray; Biological: Allergen

INTERVENTIONS:
Drug: Nasaleze Spray — Subjects are treated with over the counter Nasaleze cellulose powder nasal spray then challenged with allergen
  Arms: Nasaleze spray
Other: Placebo spray — Subjects are treated with placebo nasal spray then challenged with allergen
  Arms: Placebo spray
Biological: Allergen — Subjects are challenged with grass or ragweed allergen after treatment with Nasaleze or placebo

SUMMARY:
The objectives of this protocol are:

1. to confirm the inhibitory effect of Nasaleze on the immediate response to nasal challenge with antigen, and
2. to show that inhibition of the immediate response to nasal challenge with antigen by Nasaleze inhibits subsequent inflammatory events.

ELIGIBILITY:
Inclusion Criteria

1. Males and females between 18 and 45 years of age.
2. History of grass and/or ragweed allergic rhinitis.
3. Positive skin test to grass and/or ragweed antigen.
4. Positive response to screening nasal challenge.

Exclusion Criteria:

1. Physical signs or symptoms suggestive of renal, hepatic or cardiovascular disease.
2. Pregnant or lactating women.
3. Upper respiratory infection within 14 days of study start.
4. FEV1<80% of predicted at screening for subjects with history of mild asthma.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nasaleze Spray, Then Placebo Spray: This group first received Nasaleze spray 1 puff via "spray device" in each nostril 3 times daily for 1 week followed by allergen (either grass or ragweed) challenge, then after a 1 week washout received placebo spray 1 puff via "spray device" in each nostril 3 times daily for 1 week followed by allergen challenge
- Placebo Spray, Then Nasaleze Spray: This group first received Placebo spray 1 puff via "spray device" in each nostril 3 times daily for 1 week followed by allergen (grass or ragweed) challenge, followed by a 1 week washout and then received Nasaleze spray 1 puff via "spray device" in each nostril 3 times daily for 1 week followed by allergen challenge
Period: Study Period 1
Arm/Group | Nasaleze Spray, Then Placebo Spray | Placebo Spray, Then Nasaleze Spray
Started | 7 | 7
Completed | 7 | 6
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Washout
Arm/Group | Nasaleze Spray, Then Placebo Spray | Placebo Spray, Then Nasaleze Spray
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: Study Period 2
Arm/Group | Nasaleze Spray, Then Placebo Spray | Placebo Spray, Then Nasaleze Spray
Started | 7 | 6
Completed | 7 | 5
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Spray, Then Nasaleze Spray: This group first received placebo spray 1 puff via "spray device" in each nostril 3 times daily for 1 week followed by allergen (either grass or ragweed) challenge, then after a 1 week washout received Nasaleze spray 1 puff via "spray device" in each nostril 3 times daily for 1 week followed by allergen challenge
- Total: Total of all reporting groups
Arm/Group | Nasaleze Spray, Then Placebo Spray | Placebo Spray, Then Nasaleze Spray | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.6 (8.6) | 28.0 (7.5) | 25.8 (8.1)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Nasal Symptom Score After Nasal Challenge With Allergen Versus Diluent
Description: Change in total nasal symptom score after nasal challenges (the change is calculated as the total nasal symptom score after allergen challenge - total nasal symptom score after diluent challenge) on the second of two days of nasal challenges following one week of pretreatment with Nasaleze or placebo. The nasal symptoms included number of sneezes, symptoms of runny and stuffy nose (separately for each nostril), and itchy nose/throat symptoms. Individual symptoms were score on a scale from 0-3 (0=no symptoms, 1=mild, 2=moderate, 3=severe). The maximum total nasal symptom score possible was 15 with higher scores indicating worse symptoms.
Time Frame: Day 2 after one week pretreatment with Nasaleze or placebo.
Population: The analysis population includes the 12 participants who completed the study.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Nasaleze Spray | Placebo Spray
Number analyzed (Participants) | 12 | 12
units on a scale | 5.5 [1 to 13] | 5.5 [1 to 13]
Statistical Analysis 1: Comparison: Nasaleze Spray vs Placebo Spray; Test type: Superiority or Other; p = 0.8, Wilcoxon signed-rank test

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Nasaleze Spray | Placebo Spray
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes